

### TRIAL STATISTICAL ANALYSIS PLAN

c38727127-02

**BI Trial No.:** 1381.2

**Title:** An open label, Phase I dose-finding study of BI 754111 in

combination with BI 754091 in patients with advanced solid cancers

followed by expansion cohorts at the selected dose of the

combination in patients with non-small cell lung cancer and other

solid tumours

**Including Protocol Amendment 8** 

Investigational Products:

BI 754111 and BI 754091

Responsible trial statistician:

Phone:

Date of statistical

18 APR 2022 SIGNED

analysis plan:

**Version:** Final

**** 

Proprietary confidential information

© 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

TSAP for BI Trial No: 1381.2 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| 1. | TABLE OF CONTENTS | |
|---|---|---|
| TITLE PA | AGE | 1 |
| 1. | TABLE OF CONTENTS | 2 |
| LIST OF | ΓABLES | 4 |
| 2. | LIST OF ABBREVIATIONS | 5 |
| 3. | INTRODUCTION | 7 |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY | 8 |
| 5.<br>5.1<br>5.2<br>5.2.1<br>5.2.2 | ENDPOINTS | 9<br>9<br>9 |
| 6. | GENERAL ANALYSIS DEFINITIONS | |
| 6.1 | TREATMENTS | 3 |
| 6.2<br>6.3 | IMPORTANT PROTOCOL DEVIATIONS | |
| 6.5 | POOLING OF CENTRES1 | |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | |
| 6.7 | BASELINE, TIME WINDOWS AND CALCULATED VISITS1 | |
| 7. | PLANNED ANALYSIS | |
| 7.1 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS2 | |
| 7.2<br>7.3 | CONCOMITANT DISEASES AND MEDICATION2 TREATMENT COMPLIANCE | |
| 7.3 | PRIMARY ENDPOINTS | |
| 7.5 | SECONDARY ENDPOINTS | |
| 7.5.1 | Key secondary endpoint | |
| 7.5.2 | Other secondary endpoints | |
| 7.5.2.1 | Other secondary endpoints in Part I | |
| 7.5.2.2 | Other secondary endpoints in Part II | |
| 7.7 | EXTENT OF EXPOSURE | |
| 7.8 | SAFETY ANALYSIS | |
| 7.8.1 | Adverse events3 | 6 |

| <b>Boehringer Ingelheim</b> |
|------------------------------|
| TSAP for RI Trial No. 1391 2 |

### c38727127-02 

TSAP for BI Trial No: 1381.2 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| - | | - |
|---------|------------------------------------|----------------|
| 7.8.2 | Laboratory data | 36 |
| 7.8.2.1 | Analysis | |
| 7.8.2.2 | Classification of laboratory tests | |
| 7.8.3 | Vital signs | 41 |
| 7.8.4 | ECG | |
| 7.8.5 | Others | 41 |
| 8. | REFERENCES | 43 |
| 10. | HISTORY TABLE | 45 |
| IU. | IIISIUNI IADLE | <del>4</del> 3 |

TSAP for BI Trial No: 1381.2 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# LIST OF TABLES

| Table 6.1: 1 | Definition of analyzing treatment periods for safety analysis |
|---|---|
| Table 6.2: 1 | Important protocol deviations |
| Table 6.7: 1 | Nominal time points and windows for imaging |
| Table 6.7: 2 | Calculated visits, nominal time points and windows for laboratory assessments |
| | in Phase Ia21 |
| Table 6.7: 3 | Calculated visits, nominal time points and windows for laboratory assessments |
| | in Phase Ia |
| Table 7.4: 1 | Details of confirmed best overall response derivation rules |
| Table 7.5.2.2: | 1 Censoring rules for duration of objective response according to RECIST v1.1 |
| Table 7.5.2.2: | 3 Censoring rules for progression-free survival according to RECIST v1.130 |
| Table 7.8.2.2: | Primary Laboratory tests <sup>1</sup> |
| Table 7.8.2.2: | 2 Secondary Laboratory tests <sup>1</sup> |
| Table 7.8.2.2: | 3 Diagnostic Laboratory tests <sup>1</sup> |
| Table 7.8.2.2: | 4 Laboratory tests that will not be analyzed |
| Table 10: 1 | History table |

TSAP for BI Trial No: 1381.2 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 2. LIST OF ABBREVIATIONS

Include a list of all abbreviations used in the TSAP

| Таша | Definition / description |
|---|---|
| Term | Definition / description |
| ATC | Anatomical Therapeutic Chemical |
| AE<br>DI DM | Adverse event |
| BLRM | Bayesian logistic regression model |
| BOR | Best overall response |
| CR | Complete Response |
| CTC | Common Terminology Criteria |
| CT | Concomitant therapy |
| CTP | Clinical Trial Protocol |
| CTR | Clinical Trial Report |
| DBL | Data base lock |
| DC | Dendritic Cells |
| DLT | Dose limiting toxicity |
| DM&SM | Boehringer Ingelheim Data Management and Statistics Manual |
| DRA | Drug Regulatory Affairs |
| DMG | Dictionary Maintenance Group |
| EMA | European Medicines Agency |
| EOT | End of treatment |
| ICH | International Conference on Harmonization |
| irAE | Immune-related Adverse Event |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MQRM | Medical Quality Review Meeting |
| MTD | Maximum tolerated dose |
| O*C | Oracle Clinical |
| OR | Overall response |
| PK | Pharmacokinetics |
| PSTAT | Project Statistician |
| PT | Preferred term |
| PD | Progression of disease |
| PD | Protocol deviation |
| Q1 | Lower quartile |
| Q3 | Upper quartile |
| (i)RECIST | (immuntherapeutics) Response Evaluation Criteria in Solid Tumours |
| RPM | Report planning meeting |
| SA | Statistical analysis |
| SD | Stable Disease |
| StD | Standard deviation |
| SMQ | Standardized MedDRA query |
| SOC | System organ class |
| TESS | Treatment emergent signs and symptoms |
| ToC | Table of contents |
| TMW | Trial Medical Writer |

# **Boehringer Ingelheim**

c38727127-02 TSAP for BI Trial No: 1381.2 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TS Treated Set

Trial statistical analysis plan World Health Organization TSAP WHO

### 3. INTRODUCTION

As per ICH E9 [1], the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This TSAP assumes familiarity with the Clinical Trial Protocol (CTP), including Protocol Amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomization.

Phoenix TM WinNonlin® version 8.1 will be used for PK analyses. SAS® Version 9.4 or a newer version will be used for PK and all other analyses.

TSAP for BI Trial No: 1381.2 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

NA

#### 5. ENDPOINTS

#### 5.1 PRIMARY ENDPOINTS

The primary endpoint of Part I (dose escalation) of the trial is the:

- Maximum tolerated dose (MTD) of the BI 754111 plus BI 754091 combination
- Number of patients experiencing Dose Limiting Toxicities (DLTs) during the combination MTD evaluation period (first cycle of BI 754111 plus BI 754091 combination therapy) in patients with solid tumours.

The primary endpoint of Part II (dose expansion cohorts) of the trial is:

• Confirmed objective Response (OR), defined as the best overall response of confirmed complete response (CR) or partial response (PR) according to RECIST v. 1.1 assessed by the Investigator, where the best overall response is the best time point response recorded from the first administration of BI 754091 until the earliest of disease progression according to RECIST v1.1, death or last evaluable tumor assessment before start of subsequent anti-cancer therapy, loss to follow- up or withdrawal of consent.

#### 5.2 SECONDARY ENDPOINTS

### 5.2.1 Key secondary endpoints

No key secondary endpoints specified in CTP

### 5.2.2 Secondary endpoints

The secondary endpoints of Part I (dose escalation) of the trial are the following:

- PK parameters to be calculated for BI 754111 after single and multiple doses of BI 754111 in combination with BI 754091, and also for BI 754091 after single and multiple doses of combination therapy include:
  - C<sub>max</sub>: maximum measured concentration of BI 754111/BI 754091 in plasma
  - AUC<sub>0-504</sub>: area under the concentration-time curve of BI 754111 / BI 754091 in plasma over the time interval from 0 to 504 hours
- Number of patients experiencing DLTs from start of treatment until end of treatment (in all cycles)
- OR for patients with solid tumours: confirmed CR and PR according to RECIST Version 1.1 as assessed by the Investigator until the earliest of disease progression, death or last evaluable tumor assessment before start of subsequent anti-cancer therapy, loss to follow- up or withdrawal of consent.

The secondary endpoints of Part II (dose expansion) of the trial are the following:

- Duration of response is the duration from the date of first documented PR or CR according to RECIST Version 1.1 as assessed by the Investigator to the date of PD, up until anti-cancer therapy, or death
- Disease control (CR, PR, or SD according to RECIST Version 1.1) as assessed by the Investigator

TSAP for BI Trial No: 1381.2 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Progression-free survival (PFS) is the duration from the date of first treatment to the date of PD, up until anti-cancer therapy, or death
- Number of patients experiencing DLTs from start of treatment until end of treatment



Boehringer Ingelheim
TSAP for BI Trial No: 1381.2
Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TSAP for BI Trial No: 1381.2 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 6. GENERAL ANALYSIS DEFINITIONS

#### 6.1 TREATMENTS

In this Phase I trial, treatments are not randomized. Different dose levels of BI 754091 / BI 754111 will arise in Part I and there is only one dose level in Part II.

For Part I, the initial trial medication (*i.e.* dose level) assigned at the beginning of the first treatment cycle will be used as label of the analysing treatment.

Table 6.1: 1 Definition of analyzing treatment periods for safety analysis

| <b>Analysing Treatment</b> | Start Date | Stop Date |
|---|---|---|
| Period | | |
| Screening | Date of informed consent | Date/Time of the first |
| | | administration of trial |
| | | treatment |
| On-treatment | Date/Time of the first | Date of the last |
| | administration of trial treatment | administration of trial |
| | | treatment + 30 days (residual |
| | | effect period) |
| Follow-up | Date of the last administration of | Date of the last per protocol |
| | trial treatment + 31 days | visit |

Note: a 30-day residual effect period (REP) is defined for this trial.

For safety analyses, adverse events (AEs) will be classified to one of the following time periods: "Screening", "On-treatment" or "Follow-up". This will be applied for all adverse events. It is indicated in CTP Section 5.3.6.8.1 that the residual effect period of this trial is 30 days, and thus AE reported within 30 days of the last trial medication will be considered on treatment. Detailed rules for assigning AEs to these time periods are listed below:

- If the date of informed consent ≤ AE onset date < date/time of first administration of BI 754091 or BI 754111, then the AE is assigned to "Screening"
- If date/time of first administration of BI 754091 or BI 754111 ≤ AE onset date ≤ date of last administration of BI 754091 or BI 754111 + 30 days, then the AE is assigned to "On-treatment"
- If AE onset date > date of last administration of BI 754091 or BI 754111 + 30 days, then the AE is assigned to "Follow-up"

### 6.2 IMPORTANT PROTOCOL DEVIATIONS

According to [2] important safety protocol deviations (PDs) are those that potentially affect the rights or safety of study subjects. Important protocol deviations (IPDs) are those that can potentially influence the primary outcome measure(s) for the respective patients in a way that is neither negligible nor in accordance with the study objectives.

TSAP for BI Trial No: 1381.2 
Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

No per protocol set is defined for this phase I trial, but patients with IPDs will be identified and reported in the clinical trial report (CTR). Potential IPDs are defined in Table 6.2: 1. The final list of IPDs will be confirmed at the last report planning meeting (RPM) before data base lock (DBL).

Table 6.2: 1 Important protocol deviations

| Cate<br>Cod | egory / | Description | Comment / Example | Excluded from | Automatic/<br>Manual |
|---|---|---|---|---|---|
| A | | Entrance criteria not met | | 110111 | |
| | A1.1 | Patient < 18 years of age<br>at the time of signature of<br>ICF | Inclusion criterion (IN) 2 not met | None | Automatic |
| | A1.2 | (Dose escalation part) Patients without a confirmed diagnosis of advanced, unresectable, and/or metastatic solid tumours or any requirements of measureable disease / previous treatment status not met | IN 3 not met | None | Automatic |
| | A1.3 | (Dose expansion part) Patients without measurable disease per RECIST v1.1 criteria, or without at least 1 tumour lesion amenable to biopsy, or not medically fit and willing to undergo a biopsy before first treatment and, unless clinically contraindicated, after 6 weeks on therapy, or with any of the other cohort-specific requirements not met | IN 4 not met | None | Automatic |
| | A1.4 | ECOG score > 1 | IN 5 not met | None | Automatic |
| | A1.5 | Women of child-bearing potential and men able to father a child must be ready and able to use highly effective methods of birth control. | IN 7 not met | None | Automatic |
| | A2 | Exclusion criteria not met | | | |
| | A2.1 | Major surgery performed<br>within 12 weeks prior to<br>first trial treatment or<br>planned within 12 months<br>after screening | Exclusion criterion (EX) 1 met | None | Automatic |

TSAP for BI Trial No: 1381.2 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Category /<br>Code | Description | Comment / Example | Excluded from | Automatic/<br>Manual |
|---|---|---|---|---|
| A2.2 | Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial | EX 2 met | None | Automatic |
| A2.3 | Previous enrolment in this trial | EX 3 met | None | Automatic |
| A2.4 | Use of investigational or<br>anti-tumour treatment<br>within 4 weeks or 5 half-<br>life periods (whichever is<br>shorter) prior to the<br>initiation of trial treatment | EX 4 met | None | Automatic |
| A2.5 | Any unresolved toxicities from prior therapy greater than CTCAE Grade 1 at the time of starting study treatment with exception of alopecia and Grade 2 neuropathy due to prior platinum-based therapy | EX 5 met | None | Automatic |
| A2.6 | Prior treatment with anti-<br>LAG-3 agents | EX 6 met | None | Automatic |
| A2.7 | Patients with NSCLC that<br>has epidermal growth<br>factor receptor (EGFR)<br>mutations or anaplastic<br>lymphoma kinase (ALK)<br>rearrangements | EX 7 met | None | Automatic |
| A2.8 | Presence of other active invasive cancers others than the one treated in this trial, with the exception of resected/ablated basal or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix, or other local tumours considered cured by local treatment | EX 8 met | None | Automatic |
| A2.9 | Untreated brain<br>metastasis(es) that may be<br>considered active | EX 9 met | None | Automatic |
| A2.10 | Inadequate organ function or bone marrow reserve as demonstrated by the laboratory values in CTP Table 3.3.3:1 | EX 10 met | None | Automatic |
| A2.11 | Any of the following cardiac criteria specified in CTP Exclusion criterion 11 | EX 11 met | None | Automatic |

TSAP for BI Trial No: 1381.2 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Category /<br>Code | Description | Comment / Example | Excluded from | Automatic/<br>Manual |
|---|---|---|---|---|
| A2.12 | History of pneumonitis | EX 12 met | None | Automatic |
| 112.12 | with in the last 5 years | En 12 met | Trone | latomatic |
| A2.13 | History of severe | EX 13 met | None | Automatic |
| | hypersensitivity reactions | | | |
| | to other mAbs | | | |
| A2.14 | Immunosuppressive | EX 14 met | None | Automatic |
| | corticosteroid doses (>10 | | | |
| | mg prednisone daily or | | | |
| | equivalent) within 4 weeks | | | |
| | prior to the first dose of | | | |
| 1015 | study treatment | DY 15 | 2.7 | |
| A2.15 | Active autoimmune | EX 15 met | None | Automatic |
| | disease or a documented history of autoimmune | | | |
| | disease, except vitiligo or | | | |
| | resolved childhood | | | |
| | asthma/atopy | | | |
| A2.16 | Active infection requiring | EX 16 met | None | Automatic |
| | systemic treatment at start | | | |
| | of treatment in this trial | | | |
| A2.17 | Known history of human | EX 17 met | None | Automatic |
| | immunodeficiency virus | | | |
| | infection or active | | | |
| | hepatitis B or C virus | | | |
| 42.10 | infection | EV 10 | NT. | A |
| A2.18 | Interstitial lung disease Informed consent | EX 18 met | None | Automatic |
| B1 | Informed consent not | Inclusion criteria 1 not met | Treated Set | Automatic |
| D1 | available/not done | merasion effecta 1 not met | Treated Set | ratomatic |
| B2 | Informed consent too late | Informed consent obtained | None | Automatic |
| | | later than the initiation of | | |
| | | treatment | | |
| 7 | Trial medication | | | |
| C1.1 | Non-compliance with BI | Incorrect trial medication dose | None | Automatic and |
| | 754091 or BI 754111 per | taken or wrong dose schedule; | | manual |
| | protocol | (infusion time, program) | | |
| | | decision at MQRM | | |
| C1.2 | Discontinuation of trial | Decision at MQRM | None | Automatic and |
| | medication not following | | | manual |
| | the protocol | | | |
| ) | Concomitant medication | | | |
| D1.1 | Prohibited medication use | Review concomitant | None | Manual |
| | | medications for prohibited | | |
| | | medication use; also refer to | | |
| D . | G, 1 G 'M | Section 4.2.2.2 of the protocol | | |
| E | Study Specific | A 1 -: 4: - C | TDD | N / 1 |
| E1 | Incorrect study procedures | Any deviation from protocol | TBD | Manual |
| | performed. | not defined above deemed important to document in | | |
| | | study report by trial team. | | |

**Note:** MQRM – Medical and Quality Review Meeting; TBD – to be determined

#### 6.3 SUBJECT SETS ANALYSED

#### **Screened Set:**

This patient set includes all patients who have signed the informed consent. The screened set will be used for patient disposition tables.

#### **Treated Set (TS):**

This patient set includes all patients who were documented to have received at least one dose of BI 754091 or BI 754111. The TS is used for both efficacy analysis, safety analyses and biomarker analysis.

### MTD set:

This patient set includes all patients enrolled in Part I who were not replaced within the MTD evaluation period. Patients who were replaced during the MTD evaluation period will not be considered for MTD determination.

### PK Analysis Set (PKS):

This patient set includes all patients in the TS who provide at least one evaluable observation for at least one PK endpoint and no PK relevant protocol violation. PKS will be used for all pharmacokinetic analyses.



#### 6.5 POOLING OF CENTRES

This section is not applicable because centre/country is not included in the statistical analyses.

#### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

No imputation will be performed on missing efficacy data. No other imputations will be performed on missing data although every effort will be made to obtain complete information on all AEs, with particular emphasis on potential DLTs.

Missing or incomplete AE dates are imputed according to BI standards (see "Handling of missing and incomplete AE dates") [3].

Missing data and outliers of PK data are handled according to Boehringer internal SOPs.

In general, missing data not discussed in (3) and BI standards will not be imputed unless required for the following analyses and definitions. Then the rules as described below apply.

#### 1) Partial date for Time from First Diagnosis

If date is partial, which is allowed, then imputation will be based on below logic:

• if missing day, then imputation will use the first day of the month;

- if missing both day and month then imputation will use January 1<sup>st</sup>;
- if missing completely, then report to DM for querying the site. If the date is completely missing at the site, no imputation will be made.

### 2) Partial Start Dates of Duration of Chemotherapy or Prior Radiation

- If day is missing, then imputation will use the first day of the month;
- If month and day are missing, imputation will use January 1<sup>st</sup>.

### 3) Partial End Dates of Duration of Chemotherapy or Prior Radiation

- If day is missing, then imputation will use the later of last day of the month and the available start date;
- If month and day are missing, imputation will use the later of last day of the year and the available start date.

# 4) Partial or missing start date of subsequent anti-cancer therapy/subsequent radiotherapy

If the day of the start date of subsequent systemic therapy/subsequent radiotherapy is missing, then the 1<sup>st</sup> of the month will be imputed unless this leads to a date before the stop date of study medication. In this case the stop date of study medication +1 day will be imputed.

If day and month, or day and month and year are missing, it will be distinguished whether the start date of subsequent systemic therapy/subsequent radiotherapy is required for censoring of PFS or for other descriptive statistics:

- For censoring of PFS or DoR: If only the year is reported, the 1<sup>st</sup> of January of this year will be imputed unless this leads to a date before the stop date of study medication. In this case the stop date of study medication +1 day will be imputed. In case of a completely missing start date of subsequent anti-cancer therapy/subsequent radiotherapy and the patient did not have any post-baseline tumour assessment or did not progress or die, the PFS of this patient will be censored at the day of first administration of BI 754091 or BI 754111. Additionally, all imputed start dates of subsequent anti-cancer therapy/subsequent radiotherapy should be before the death date, if available.
- <u>For descriptive statistics:</u> Dates will not be imputed if more than only the day of the date is missing.

#### 5) Partial death date / end of study date

If the day of the death/end of study date is missing, then the 1<sup>st</sup> of the month will be imputed.

### 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

Unless otherwise specified baseline is defined as the time point closest to but prior to the first administration of any study medication. If no time is specified and the date is the same as the first administration date, then it will still be considered baseline if not specified otherwise. If there is no measurement earlier than the first administration of study medication, then no baseline will be derived.

Study day will be calculated relative to the date of the first administration of study drug. The day prior to first administration of study drug will be 'Day -1' and the day of first administration of study drug will be 'Day 1'; therefore 'Day 0' will not exist.

### Imaging time windows:

Time windows and visits will be calculated to determine the planned day of tumour measurement and response status, based on the protocol-specified tumour imaging schedule.

For the presentation of tumour response data which will follow a calculated visit approach based on the protocol specified tumour imaging schedule. Imaging will be performed at screening and every 6 weeks after BI 754091 infusion (i.e. Week 6, 12, 18 ...etc.), then every 9 weeks after 6 months of treatment; image data will be slotted to Week 6, 12, 18 etc. based on their relative day (from start of treatment) and using a  $\pm 3$  week window (images taken in the first 3 weeks from start of treatment will be assigned to Week 6). If two or more images for a patient are assigned to one interval then the last assessment will be used to ensure progressive disease is not missed.

In order to identify whether consecutive imaging time points are missing for a given patient, a nominal time point (i.e. Week 6, 12, 18 ... etc.) will be assigned to each and every image. This is achieved by creating windows for every radiological response assessment. These windows are defined in <u>Table 6.7: 1</u>.

| Table 6.7: 1 | Nominal time | points and | windows | for | imaging |
|--------------|--------------|------------|---------|-----|---------|

| Nominal time point (weeks from start of study medication) | Due date of scans (days)* | Window (days) |
|---|---|---|
| 6 | 43 | 1 to ≤ 64 |
| 12 | 85 | 65 to ≤ 106 |
| 18 | 127 | $107 \text{ to} \le 148$ |
| 24 | 169 | 149 to $\leq$ 200 |

<sup>\*</sup> The date of the first dose of study medication is Day 1

Table 6.7: 2 Nominal time points and windows for imaging (cont.)

| Nominal time point (weeks from start of study medication) | Due date of scans (days)* | Window (days) |
|---|---|---|
| 33 | 232 | $201 \text{ to } \le 263$ |
| 42 | 295 | 264 to ≤ 326 |
| 51 | 358 | $327 \text{ to} \le 389$ |
| Etc., 9 week interval | Etc. | Etc. |

<sup>\*</sup> The date of the first dose of study medication is Day 1

If a patient does not have an image in one of the windows described above, he/she will be said to have missed an assessment for that time point.

### Laboratory values:

Baseline is defined as the latest time point before the very first administration of any study medication. For laboratories where not only the examination date but also time are recorded, examination time has to be taken into account when defining baseline. That is, a laboratory value on the same date as the first administration of study medication is considered as baseline value if and only if the time of laboratory assessment is before or the same as the time of first study drug administration.

If any of these times is missing and the date of laboratory assessment is equal to the date of first administration of study medication, then the laboratory assessment will be considered as according to protocol, i.e. as prior to first study medication.

### Laboratory time windows:

Time windows and visits will be calculated to determine the planned day of laboratory assessment, based on the protocol-specified laboratory assessment schedule.

For the presentation of a descriptive summary analysis over time for a laboratory parameter the laboratory data will be displayed by calculated visit instead of actual visit reported to ensure a common handling of all laboratory assessments and to account for unscheduled visits representing a repeated laboratory measurement. As Phase Ia and Phase Ib have a different laboratory assessment schedule, the time windows for the calculated visits will be different for Phase Ia and Phase Ib.

TSAP for BI Trial No: 1381.2 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Calculated visits, nominal time points and windows for laboratory assessments in Phase Ia

| Calculated visit | Nominal time point (day from start of study medication)* | Window (days) |
|---|---|---|
| Cycle 1 Day 1 | 1 | 1 to ≤ 4 |
| Cycle 1 Day 8 | 8 | 5 to ≤ 11 |
| Cycle 1 Day 15 | 15 | 12 to ≤ 18 |
| Cycel 2 Day 1 | 22 | 19 to ≤ 32 |
| Cycle 3 Day 1 | 43 | 33 to ≤ 53 |
| Cycle 4 Day 1 | 64 | 54 to ≤ 74 |
| Etc., 21 days interval | Etc. | Etc. |

<sup>\*</sup> The date of the first dose of study medication is Day 1

Table 6.7: 3 Calculated visits, nominal time points and windows for laboratory assessments in Phase Ia

| Calculated visit | Nominal time point (days from start of study medication)* | Window (days) |
|---|---|---|
| Cycle 1 Day 1 | 1 | 1 to ≤ 11 |
| Cycel 2 Day 1 | 22 | 12 to ≤ 32 |
| Cycle 3 Day 1 | 43 | 33 to ≤ 53 |
| Cycle 4 Day 1 | 64 | 54 to ≤ 74 |
| Cycel 5 Day 1 | 85 | 75 to ≤ 95 |
| Cycle 6 Day 1 | 106 | 96 to ≤ 116 |
| Cycle 7 Day 1 | 127 | $117 \text{ to} \leq 137$ |
| Cycel 8 Day 1 | 148 | $138 \text{ to} \le 158$ |
| Cycle 9 Day 1 | 169 | 159 to $\leq$ 179 |
| Cycle 12 Day 1 | 232 | $180 \text{ to} \le 1263$ |
| Cycel 15 Day 1 | 295 | 264 to ≤ 326 |
| Cycle 18 Day 1 | 358 | $327 \text{ to} \le 389$ |
| Etc., 21 days interval | Etc. | Etc. |

<sup>\*</sup> The date of the first dose of study medication is Day 1

### Biomarker time windows:

The time windows used for biomarker analysis are defined as follows.

### Cytokine / flow cytometry:

C1D1 (BL): before 1st treatment (1T)

C1D2: 24h post 1T +/-18 h C1D8: 168 h post 1T +/- 48 h C1D15: 336 h post 1T +/- 48 h

C2D1: before 2nd treatment (2T) -24 h

C2D2: 24h post 2T +/-18 h C2D8: 168h post 2T +/- 48 h

C3D1: before 3rd treatment (3T) -24 h

### **Boehringer Ingelheim** TSAP for BI Trial No: 1381.2

c38727127-02

TSAP for BI Trial No: 1381.2 
Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

C4D1: before 4th treatment (4T) -24 h

C4D2: 24h post 4T +/-18 h C4D8: 168h post 4T +/- 48 h

C5D1: before 5th treatment (5T) -24 h

Biopsies (Immunohistochemistry, RNAseq):

C1D1: before 1st treatment (1T)

C3D1: 1008 h post 1st Treatment +/- 168 h

### 7. PLANNED ANALYSIS

For End-Of-Text tables, the set of summary statistics is: N / Mean / Standard deviation (StD) / Min / Median / Max.

For tables that are provided for endpoints with some extreme data, median, quartiles and percentiles should be preferred to Mean, StD, Min and Max.

For time-to-event analysis tables the set of statistics is: number of patients [N(%)], number of patients with event [N(%)], <time to event> [months] followed by P25 (25<sup>th</sup> percentile), median, P75 (75<sup>th</sup> percentile) and number of patients censored [N(%)]. If not specified otherwise the duration as well as the time to event will be displayed in months.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%) relative to the respective treatment group (unless otherwise specified, all patients in the respective patient set whether they have non-missing values or not). Percentages will be rounded to one decimal place. The category missing will be displayed only if there are actually missing values.

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Descriptive statistics are planned for demographic characteristics, disease history, prior therapies, medical history, alcohol and tobacco use, baseline ECOG PS, and baseline disease assessment.

### 7.2 CONCOMITANT DISEASES AND MEDICATION

Only descriptive statistics are planned for this section of the report. Concomitant diseases will be coded similarly as adverse events based on the most current Medical Dictionary for Regulatory Activities (MedDRA) version. Concomitant therapies (CTs) will be coded according to World Health Organization (WHO) Drug Dictionary (actual version). CTs will be classified according to the Anatomical Therapeutic Chemical (ATC) classification system. The third ATC level will be used to categorize CTs by therapy type. In situations where a medical product may be used for more than one equally important indication, there are often several classification alternatives. As appropriate, patients receiving CTs with more than one possible ATC level 3 category will be counted more than once. Footnotes will clarify this possible double counting in tables.

#### 7.3 TREATMENT COMPLIANCE

Not applicable in this study.

### 7.4 PRIMARY ENDPOINTS

In order to identify the MTD and the recommended dose for Part II, the number of patients with DLTs at each dose level during Part I (first three weeks) must be presented. Patients who discontinue during the first treatment course for reasons other than a DLT will be excluded from the determination of the MTD.

The analysis of the MTD is based on a BLRM guided by the escalation with overdose control principle. The MTD is defined as the highest dose for a given schedule that is expected to cause less than 25% risk of the true DLT rate being above or equal to 33% during the MTD evaluation period. Estimation of the MTD during the dose escalation phase of the study will be based upon the estimation of the posterior probability of the incidence of DLT in toxicity categories during the MTD evaluation period for all evaluable patients. The model to be used is specified in CTP Section 7.

In addition, the number of patients with DLTs that occurred during Part I and Part II will be summarized at each dose level. The BLRM will be rerun to re-evaluate the MTD and RP2D together with all relevant data collected during Part II.

For Part II, OR according to RECIST Version 1.1 will be summarized descriptively with exact 95% Clopper-Pearson CIs. Response data collected after the EOT, after PD, or the start of subsequent anti-cancer therapy will not be used. This applies to other endpoints based on the response data. Confirmed best overall response (BOR) will be derived according to the following derivation rules:

Table 7.4: 1 Details of confirmed best overall response derivation rules

| Overall response (time point 1) | Overall response (>=28 days from time point 1) | Confirmed BOR |
|---|---|---|
| CR | CR | CR |
| CR | PD | SD as long as >=39 days, otherwise, PD |
| CR | NE/Missing | SD as long as >=39 days, otherwise, NE |
| PR | CR | PR |
| PR | PR | PR |
| PR | SD | SD as long as >=39 days, otherwise, PD |
| PR | PD | SD as long as >=39 days, otherwise, PD |
| PR/SD | NE/Missing | SD as long as >=39 days, otherwise, NE |

NE: not evaluable

- If CR or PR: Look at all subsequent visits, if there is another CR or PR >=28 days and no more than one missing visit (defined by time window Table 6.7.1) in between then the patient has a confirmed response. If there is not another CR or PR >=28 days and/or more than one missing visit between the two responses, then the patient can be a confirmed SD if the CR or PR is >=39 days from start of combination therapy.
- If SD: To be confirmed SD, the measurement must have been taken >=39 days from start of combination therapy (only one reading is necessary).
- Additional details are provided in Table 7.4: 1.

#### 7.5 SECONDARY ENDPOINTS

### 7.5.1 Key secondary endpoint

This section is not applicable as no key secondary endpoint has been defined in protocol.

### 7.5.2 Other secondary endpoints

### 7.5.2.1 Other secondary endpoints in Part I

PK parameters evaluated after the single and after multiple administrations of BI 754111 in combination with BI 754091, and also for BI 754091 after single and multiple doses of combination therapy

The PK parameters will be evaluated using noncompartmental analysis methods according to 001-MCS-36-476 [4]. Tables and figures for concentration values and PK parameters will be created according to Boehringer internal SOPs.

Descriptive statistics will be calculated for all concentration time points and PK parameters. The following descriptive statistics will be calculated for BI 754111 and BI 754091 concentrations and for PK parameters: N, arithmetic mean, standard deviation, minimum, median, maximum, tenth percentile (P10), Q1, Q3, ninetieth percentile (P90), arithmetic coefficient of variation, geometric mean, and geometric coefficient of variation.

Treated and evaluable patients will be included in the PK analysis. A patient is considered not evaluable if the patient had an important protocol violation relevant to the evaluation of PK or had insufficient PK data. Non evaluable patients will be listed with their individual PK parameters, but such data will not be included when calculating descriptive statistics. If the data suggest a PK / PD relationship of special parameters (e.g. PK vs. RO), a detailed analysis may be performed and documented in a separate report.

Number of patients experiencing DLTs from the start of treatment until end of treatment

Number of patients with DLT(s) which occurred during the entire treatment period will be summarized for each dose cohort.

OR for patients with solid tumors according to RECIST Version 1.1 as assessed by the investigator

OR will be summarized descriptively with exact 95% Clopper-Pearson CIs.

### 7.5.2.2 Other secondary endpoints in Part II

Duration of response according to RECIST Version 1.1 as assessed by the Investigator

Duration of response is defined as the duration from the date of first documented PR or CR according to RECIST Version 1.1 as assessed by the Investigator to the date of PD, up until anticancer therapy, or death. Duration of response will be provided in a listing.

Duration of OR according to RECIST v1.1:

Duration of OR can only be calculated for patients with OR.

For patients with disease progression or death:

- Duration of OR [days] = date of outcome date of first assessment indicating OR + 1 For patients without disease progression or death:
  - Duration of OR (censored) [days] = date of outcome date of first assessment indicating OR + 1

Censoring rules and applicable dates of outcome for duration of OR according to RECIST v1.1 are specified in Table 7.5.2.2:1

Table 7.5.2.2:1 Censoring rules for duration of objective response according to RECIST v1.1

| Situation | Outcome<br>(event or<br>censored) | Date of outcome |
|---|---|---|
| No other anti-cancer therapy | | |
| Alive and not progressed according to RECIST v1.1, no missed radiological assessment window* | Censored | Date of last radiological assessment |
| Alive and not progressed according to RECIST v1.1, one or more consecutively missed radiological assessment window* | Censored | Date of last radiological assessment prior to missed radiological assessments |
| Progressed according to RECIST v1.1, no missed radiological assessment window* prior to progression | Event | Date of radiological assessment of progression |
| Progressed according to RECIST v1.1, one or more consecutively missed radiological assessment window* prior to progression | Censored | Date of last radiological assessment prior to missed assessments |
| Death but no progression according to RECIST v1.1, no missed radiological assessment window* prior to death | Event | Date of death |

TSAP for BI Trial No: 1381.2 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 7.5.2.2:1 Censoring rules for duration of objective response according to RECIST v1.1 (cont.)

| Situation | Outcome<br>(event or | Date of outcome |
|---|---|---|
| | censored) | |
| Death without progression according to RECIST v1.1, but one or more consecutively missed radiological assessment window* prior to death | Censored | Date of last radiological assessment prior to missed assessments |
| Initiation of subsequent anti-cancer therapy | 7 | |
| Subsequent anti-cancer therapy started before progression according to RECIST v1.1 or death, no missed radiological assessments prior to start of subsequent anti-cancer therapy | Censored | Date of last radiological assessment before initiation of subsequent anti-cancer therapy |



Censoring rules and applicable dates of outcome for duration of OR according to RECIST v1.1 are specified in Table 7.5.2.2:2.



TSAP for BI Trial No: 1381.2 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Disease control according to RECIST Version 1.1 as assessed by the Investigator

Disease control is defined as a BOR of CR, PR or SD. Disease control rates will be presented with exact 95% Clopper-Pearson CIs.

PFS

PFS [days] = date of outcome – date of first administration of any trial medication + 1. A patient has an evaluable response assessment if CR, PR, stable disease (SD), or progressive disease (PD) according to RECIST v1.1 has been assigned by the investigator. PFS will be summarized descriptively by quartiles with 95% confidence interval (based on the Greenwood's method) calculated from Kaplan-Meier estimate. Kaplan-Meier plots will also be produced. Rules to determine censoring, PFS events and applicable dates of outcome are specified in Table 7.5.2.2: 3 below.

If patients would have their radiological examinations over a number of days, (*i.e.* target lesions assessed on day x, non-target lesions assessed on day y and new lesion (if applicable) on day z), the earliest date of the multiple assessments should be considered.

Table 7.5.2.2:3 Censoring rules for progression-free survival according to RECIST v1.1

| Situation | Outcome | Date of outcome |
|---|---|---|
| No baseline radiological assessment | | |
| Patient with death on or before first planned post-baseline radiological assessment (≤ Day 64) | Event | Date of death |
| Patient without death or patient with death after first planned post-baseline radiological assessment (> Day 64) | Censored | First treatment administration |
| Without post-baseline radiological as | sessments | |
| Vital status is unknown or patient is known to be alive | Censored | First treatment administration |
| Death prior to or on the first planned post-baseline radiological assessment (≤ Day 64) | Event | Date of death |

TSAP for BI Trial No: 1381.2 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Situation | Outcome | Date of outcome |
|---|---|---|
| Death beyond the first planned post-baseline radiological assessment (> Day 64) | Censored | First treatment administration |
| With baseline and post-baseline radio | ological assessi | ments BUT no other anti-cancer therapy |
| Alive and not progressed | Censored | Date of last evaluable radiological assessment |
| Progressed, no missed radiological assessment window* prior to progression | Event | Date of radiological assessment of progression |
| Progressed, but one or more consecutively missed radiological assessment window* prior to progression | Censored | Date of last evaluable radiological assessment prior to missed assessment (or first treatment administration if no post-baseline assessment prior to missed assessment) |
| Death but no progression, no missed radiological assessment window* prior to death | Event | Date of death |
| Death without progression, but one or more consecutively missed radiological assessment window* prior to death | Censored | Date of last evaluable radiological assessment prior to missed assessments |
| Initiation of subsequent anti-cancer the | nerapy | |
| Subsequent anti-cancer therapy started before progression or death | Censored | Date of last radiological assessment before subsequent anti-cancer therapy |
| No baseline and/or post-baseline imaging and subsequent-anti cancer therapy started prior to death | Censored | First treatment administration |

<sup>\*</sup> Windows for radiological assessments are defined in Table 6.7: 1



TSAP for BI Trial No: 1381.2 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



TSAP for BI Trial No: 1381.2 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



TSAP for BI Trial No: 1381.2 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



Number of patients experiencing DLTs from start of treatment until end of treatment

Number of patients with DLT(s) which occurred during the entire treatment period will be summarized for each expansion cohort.



TSAP for BI Trial No: 1381.2 
Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



#### 7.7 **EXTENT OF EXPOSURE**

The total number of cycles initiated and the numbers of cycle initiated will be summarized descriptively for each dose cohort. Results from Part I and Part II will be presented separately.

#### 7.8 **SAFETY ANALYSIS**

All safety analyses will be performed on the TS.

Patients who were replaced within the MTD evaluation period will be excluded from the determination of the MTD but will be considered for all other safety evaluations.

#### 7.8.1 Adverse events

Unless otherwise specified, the analyses of AEs will be descriptive in nature. All analyses of AEs will be based on the number of subjects with AEs and not on the number of AEs. The reporting and analyses of AEs will follow the BI guideline [5]. AEs will be coded with the most recent version of MedDRA®. The severity of AEs will be scaled according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

Unless otherwise specified, the analysis of adverse events will be based on the concept of treatment emergent adverse events. For details on the treatment definition, see <u>Section 6.1</u>.

An overall summary of AEs will be presented with an additional entry for patients with DLT(s) and will also include the number of patients with AEs by the worst CTCAE grade.

The frequency of patients with AEs will be summarized by treatment, primary system organ class and/or preferred term, and will be sorted by the highest CTCAE grade. Separate tables will be provided for patients with:

- DLTs
- All adverse events
- Serious adverse events
- Drug-related AEs
- Drug-related serious AEs
- AEs leading to permanent discontinuation of trial treatment
- AEs leading to death
- Treatment emergent immune-related AEs (irAEs)
- irAEs through the whole trial
- Infusion-related AEs

The system organ classes will be sorted by frequency, and preferred terms will be sorted by frequency (within system organ class).

### 7.8.2 Laboratory data

The analysis of laboratory data will be descriptive in nature and will be based on BI standards [6]. The same on-treatment period as considered for the analysis of adverse events will be applied for laboratory values. Patients having at least one post-baseline laboratory value will be displayed in the descriptive analyses. Patients with missing CTCAE grade at baseline or no baseline value but with post-baseline values will be displayed in a new category "missing CTCAE grade at baseline" for those laboratory parameters where CTCAE grading is applicable. CTCAE grades for applicable laboratory parameters will be calculated according to CTCAE Version 5.0.

### 7.8.2.1 Analysis

The Laboratory tests will be classified into the following categories:

- Primary- full analysis
- Secondary- listing of possible clinically significant values
- Diagnostic- listing of all observed values
- Not analysed

The following outputs will be presented for primary laboratory tests:

- Descriptive statistics, including changes from baseline
- Frequency of patients with shifts from baseline
  - o Shifts will be defined in terms of
    - CTCAE grades will be used for laboratory tests with CTCAE grades defined
    - The upper and lower reference limits will be used for laboratory tests without CTCAE grades
- Frequency of patients with possible clinically significant abnormalities (definitions see Section 7.8.2.2)

The analysis of secondary laboratory tests will be limited to tabulation of the frequency of patients with possible clinically significant abnormalities (definitions see <u>Section 7.8.2.2</u>).

Laboratory tests classified as "diagnostic" are recorded as a follow-up to abnormalities of associated lab tests for diagnostic purposes i.e. amylase and lipase would be measured to investigate possible pancreatitis. These values will be presented in a separate listing. No other analyses will be performed

Analyses of descriptive statistics should use normalized lab values and will be displayed by calculated visit instead of actual visit reported to ensure a common handling of all laboratory assessments and to account for unscheduled visits representing a repeated laboratory measurement (see Table 6.7: 2 and Table 6.7: 3).

Analyses of frequencies of patients with potential clinical significance, analyses of shift, and liver function categories tables should use converted values.

Baseline for safety laboratory parameters will be the last available measurement before the start of study drug. Laboratory measurements taken up to 30 days after the last administration of study drug will be considered as on-treatment.

Primary laboratory test results will be presented in CTR section 15. Laboratory test that are not analysed will be listed in Appendix 16.2.8.

### Handling of CTCAE grade -1 and -9 laboratory parameters:

Generally, in case only one direction of worsening (high or low laboratory value) is specified in the CTCAE document, there is no need to examine the other direction. Therefore, for calculating the change in CTCAE grade, patients with a CTCAE grade of -9 (no CTCAE grade defined) will be automatically treated as CTCAE grade 0 for all analyses. In laboratory listings, the CTCAE grade will be displayed as -9.

There are certain parameters for which CTCAE grades can only be differentiated by taking physiological consequences into account. These laboratory values will be coded as -1. As these definitions aggregate laboratory data and adverse events or concomitant therapies no analyses based on CTCAE grades will be done. Instead standard laboratory analyses as for laboratory parameters without CTCAE grade definitions will be done.

### Corrected calcium:

The grading of hypocalcemia is based on corrected calcium as calcium can be falsely low if hypoalbuminemia is present. The following corrective calculation will be performed:

Corrected calcium (mg/dL) = Total Calcium (mg/dL) – 0.8 [Albumin (g/dL) – 4g/dL]

No correction of the reference range has to be done. The reported reference range of total calcium will be used for analyses.

Corrected calcium can be only derived at a certain time point in case both laboratory values total calcium and albumin have been reported for the patient in the same laboratory sample.

### Differential blood count:

Differential blood counts were to be measured in absolute values according to the CTP. In case a subject's differential blood count is reported in percentage, the following conversion will be applied:

Differential  $[10^9/L]$  = Differential [%] \* (White blood cell count value / 100)

The corresponding reference ranges of the converted differential blood values are not allowed to be converted like the individual laboratory measurements. The reference range is taken from the BI standard reference range definition.

#### Liver Function tests and potential Hy's Law

A listing of all liver function tests will be provided for all patients who meet the following criteria at any time:

• ALT or AST  $\ge 3x$ ULN and elevation of total bilirubin  $\ge 2x$ ULN at within +/-30 days

In addition, tables of liver function test abnormalities will be produced.

TSAP for BI Trial No: 1381.2 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7.8.2.2 Classification of laboratory tests

Primary Laboratory tests<sup>1</sup> Table 7.8.2.2: 1

| Label | Lab test name | Direction | Potential Clinical significance |
|---|---|---|---|
| | | of interest | rule |
| ALKP | Alkaline Phosphatase | High | CTCAE Grade 2 or higher <sup>4</sup> |
| BILI | Total Bilirubin | High | CTCAE Grade 2 or higher <sup>4</sup> |
| BILDIR | Direct Bilirubin | High | CTCAE Grade 2 or higher <sup>4</sup> using |
| | | | grades defined for Total Bilirubin |
| CK | Creatinine Kinase | High | $A^{2,3}$ |
| CREJIDMS | Creatinine | High | >1.5xULN and >baseline |
| | | | ambiguous CTCAE not used <sup>4</sup> |
| FT3 | Triiodothyronine, Free | Low <sup>5</sup> , | <lln <baseline="" and="" or<="" td=""></lln> |
| | | High <sup>5</sup> | >ULN and >baseline |
| | | | No CTCAE defined |
| FT4V | Thyroxine, Free | Low <sup>5</sup> , | <lln <baseline="" and="" or<="" td=""></lln> |
| | | High <sup>5</sup> | >ULN and >baseline |
| | | | No CTCAE defined |
| GLUB | Glucose | Low, High <sup>5</sup> | Low: A <sup>2,3</sup> |
| | | | High: >10mmol/L and > baseline |
| | | | No CTCAE defined |
| HGB | Hemoglobin | Low | A <sup>2,3</sup> (listed in CTCAEv5 as |
| | | | "Anemia") |
| K | Potassium | Low <sup>5</sup> , High | Low: < 3 mmol/L and <baseline< td=""></baseline<> |
| | | | High: A <sup>2,3</sup> |
| LDH | Lactate Dehydrogenase | High <sup>5</sup> | ≥ 3xULN and > baseline |
| | | | No CTCAE defined |
| LYMABS | Lymphocytes | Low | $A^{2,3}$ |
| NA | Sodium | Low <sup>5</sup> , High | High: A <sup>2,3</sup> |
| | | | Low: < 130mmol/L and < baseline |
| NEUABS | Neutrophils | Low | $A^{2,3}$ |
| PLTCT | Platelets | Low | $A^{2,3}$ |
| SGOT | Aspartate Aminotransferase | High | CTCAE Grade 2 or higher <sup>4</sup> |
| SGPT | Alanine Aminotransferase | High | CTCAE Grade 2 or higher <sup>4</sup> |
| TPONI | Troponin I | High <sup>5</sup> | >ULN and > baseline |
| | | | CTCAE based upon AE |
| TPONTULT | Troponin T | High <sup>5</sup> | >ULN and > baseline |
| | | | CTCAE based upon AE |
| TSH | Thyrotropin | Low <sup>5</sup> , | <lln <baseline="" and="" or<="" td=""></lln> |
| | | High <sup>5</sup> | >ULN and >baseline |
| | | | No CTCAE defined |
| UREAN | Blood Urea Nitrogen | High <sup>5</sup> | > 10 mmol/L and > baseline |
| | | | No CTCAE defined |
| WBC | Leukocytes | Low | $A^{2,3}$ |

<sup>&</sup>lt;sup>1</sup> Shift tables, descriptive statistics, and potential clinically significant values will be presented.

Table 7.8.2.2: 2 Secondary Laboratory tests<sup>1</sup>

| Label | Lab test name | Direction of | Potential Clinical significance |
|---|---|---|---|
| | | interest | rule |
| ALB | Albumin | Low | $A^2$ |
| CA | Calcium | Low, High | $A^2$ |
| CHOL | Cholesterol | High | $A^2$ |
| CL | Chloride | Low, High | <80 mmol/L and <baseline< td=""></baseline<> |
| | | | or |
| | | | >120 mmol/L and >baseline |
| | | | No CTCAE defined |
| CPEP | C-peptide | Low | <lln <baseline<="" and="" td=""></lln> |
| | | | No CTCAE defined |
| EOSABS | Eosinophils | High | >1.0 10**9/L and |
| | | | > baseline |
| | | | No CTCAE defined |
| P | Phosphate | Low, High | H: > 1.7 mmol/L and >baseline, |
| | | | L: < 0.7 mmol/L and <baseline< td=""></baseline<> |
| PROT | Serum Protein | Low | <lln <baseline<="" and="" td=""></lln> |
| | | | No CTCAE defined |
| TRIGL | Triglycerides | High | $A^2$ |
| UREA | Urea | High | > 1.5 x ULN and > baseline |
| | | | No CTCAE defined |
| URIC | Uric Acid | High | Females: > 600umol/L |
| | | | and >baseline |
| | | | Males: > 650umol/L |
| | | | and >baseline |
| | | | CTCAE based upon AE |

<sup>&</sup>lt;sup>1</sup> The frequencies of potential clinically significant values will be tabulated, and values that meet the criteria will be listed. No other analyses will be performed.

<sup>&</sup>lt;sup>2</sup> A= CTCAE grade 2 or greater with an increase of at least one CTCAE grade from baseline

<sup>&</sup>lt;sup>3</sup> Separate shift tables for the low and high directions, when both directions are specified. Shift tables compare baseline vs. on-treatment CTCAE grades. CTCAE grading will not consider symptoms.

<sup>&</sup>lt;sup>4</sup> CTCAE grades will not be defined for baseline values for ALKP, SGPT, SGOT, BILI (Total and Direct) and baseline and post-baseline values for CREJIDMS. Special categories are defined for shift tables.

<sup>&</sup>lt;sup>5</sup> Separate shift tables for the low and high directions, when both directions are specified. Shift tables compare baseline vs. on-treatment using the three categories 1.) below reference range, 2.) within reference range, and 3.) above reference range.

<sup>&</sup>lt;sup>2</sup> A= CTCAE grade 2 or greater with an increase of at least one CTCAE grade from baseline

<sup>&</sup>lt;sup>3</sup> CTCAE grading will not consider symptoms such as presence of bleeding or use of anticoagulation.

Table 7.8.2.2: 3 Diagnostic Laboratory tests<sup>1</sup>

| Label | Lab test name | Direction of interest | Potential Clinical significance rule |
|---|---|---|---|
| AMYL | Amylase | High | > 2x ULN and > baseline |
| LIPASE | Lipase | High | > 2x ULN and > baseline |

<sup>&</sup>lt;sup>1</sup>Values will be displayed in a listing. No other analysis will be performed.

Table 7.8.2.2: 4 Laboratory tests that will not be analyzed

| Label | Lab test name |
|---------|------------------------------|
| BASABS | Basophils |
| BICARBV | Bicarbonate |
| CKMBABS | Creatinine Kinase MB |
| HCT | Hematocrit |
| HDL | HDL Cholesterol |
| LDL | LDL Cholesterol |
| MCV | Ery. Mean Corpuscular Volume |
| MONABS | Monocytes |
| PREG | Choriogonadotropin Beta |
| RBC | Erythrocytes |
| UGLU | Urine Glucose |
| UNIT | Urine Nitrite |
| UPH | Urine pH |
| UPRO | Urine Protein |
| URBCZ | Urine Erythrocytes |
| UWBCZ | Urine Leukocytes |

### 7.8.3 Vital signs

Only descriptive statistics are planned for this section of the report.

### 7.8.4 ECG

Clinically significant abnormal ECG findings (as assessed by the investigator) will be provided in the form of patient level listing.

### **7.8.5** Others

TSAP for BI Trial No: 1381.2 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



TSAP for BI Trial No: 1381.2 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 8. **REFERENCES**

IDEA for CON.

| 1. | CPMP/ICH/363/96: "Statistical Principles for Clinical Trials", ICH Guideline Topic E9, Note For Guidance on Statistical Principles for Clinical Trials, current version. |
|---|---|
| 2. | 001-MCS-50-413: "Handling of Protocol Violations in Clinical Trials and Projects", current version; group: Study Conduct; IDEA for CON. |
| 3. | 001-MCG-156_RD-01: "Handling of missing and incomplete AE dates", current version; IDEA for CON. |
| 4. | 001-MCS 36-472: "Standards and processes for analyses performed within Clinical Pharmacokinetics/Pharmacodynamics", current version; IDEA for CON. |
| 5. | 001-MCG-156: "Handling and summarization of adverse event data for clinical trial reports and integrated summaries", current version; IDEA for CON. |
| 6 | 001-MCG-157: "Handling, Display and Analysis of Laboratory Data", current version: |

TSAP for BI Trial No: 1381.2 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies



TSAP for BI Trial No: 1381.2 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 10. HISTORY TABLE

Table 10: 1 History table

| Version | Date<br>(DD-MMM-YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| Initial | 21-JUN-17 | | None | This is the initial TSAP with necessary information for trial conduct. |
| Final | DD-MMM-19 | None This is the final TSAP | | |
| Draft 3.2 | 18-APR-22 | | 6.6 | Added imputation rules for partial dates |



### APPROVAL / SIGNATURE PAGE

Document Number: c38727127 Technical Version Number: 2.0

**Document Name:** 8-01-tsap-core-3

**Title:** An open label, Phase I dose-finding study of BI 754111 in combination with BI 754091 in patients with advanced solid cancers followed by expansion cohorts at the selected dose of the combination in patients with non-small cell lung cancer and other solid tumours

### Signatures (obtained electronically)

| Meaning of Signature | Signed by | Date Signed |
|--------------------------------|-----------|------------------------|
| Author | | 19 Apr 2022 14:19 CEST |
| Approval-Biostatistics | | 19 Apr 2022 15:19 CEST |
| Approval-Clinical Program | | 19 Apr 2022 16:20 CEST |
| Approval-Clinical Trial Leader | | 22 Apr 2022 10:54 CEST |

Boehringer IngelheimPage 2 of 2Document Number: c38727127Technical Version Number: 2.0

(Continued) Signatures (obtained electronically)

| Meaning of Signature | Signed by | <b>Date Signed</b> |
|----------------------|-----------|--------------------|
|----------------------|-----------|--------------------|